CLINICAL TRIAL: NCT06591676
Title: Translation and Cultural Adaptation of the Dysfunctional Attitude Scale (DAS) Into Urdu
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACTDAS24
Record Dates: First submitted 2024-06-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Depression; Anxiety
Keywords: DAS; CBT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial to evaluate the feasibility and acceptability of delivering a new intervention. Participants who meet the inclusion criteria will be randomly allocated to intervention or control groups in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- administration of DAS in samples of outpatients (Experimental)
  Interventions: Behavioral: Dysfunctional Attitude Scale (DAS)
- administration of DAS in samples of students (Experimental)
  Interventions: Behavioral: Dysfunctional Attitude Scale (DAS)

INTERVENTIONS:
Behavioral: Dysfunctional Attitude Scale (DAS) — Dysfunctional Attitude Scale (DAS) is a self-report scale designed to measure the presence and intensity of dysfunctional attitudes. It is widely used to assess impaired cognitive patterns associated with depression and other mental health conditions. Initially developed in English, its usefulness can be extended by translating and culturally adapting it into Urdu language.

SUMMARY:
Translate and adapt the Dysfunctional Attitude Scale (DAS) into Urdu language and establishing the psychometric properties (reliability, validity, and norms) of the translated scale

DETAILED DESCRIPTION:
the present study aims to translate and culturally adapt the Dysfunctional Attitude Scale (DAS) into Urdu language. This study aims to increase the accessibility and accuracy of clinical assessments, ultimately improving the quality of mental health care delivery and advancing research in the field of clinical psychology within Urdu-speaking communities.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 18 to 65 years At least 5 years of education Individuals with symptoms of Depression and Anxiety

-

Exclusion Criteria:

* Substance use disorder according to DSM-5 TR criteria Significant cognitive impairment (for example, profound learning disability or dementia) Active psychosis as determined by their primary care clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2024-09-08 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cultural adapatation of DAS | 12 weeks
  facilitating access and use of the DAS for Urdu-speaking patients/clients, thereby facilitating more accurate assessments of psychopathology and maladjustment.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided